CLINICAL TRIAL: NCT04350463
Title: A Phase 2, Multicenter, Open-label, Multi-cohort Study to Assess Safety and Efficacy of CC-90011 in Combination With Nivolumab in Subjects With Advanced Cancers
Brief Title: A Safety and Efficacy Study of CC-90011 in Combination With Nivolumab in Subjects With Advanced Cancers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CC-90011-ST-002; U1111-1248-8352 (Other: WHO); 2019-004194-95 (EudraCT Number)
Record Dates: First submitted 2020-03-20; First posted 2020-04-17 (Actual); Results first posted 2025-01-22 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Neoplasms
Keywords: CC-90011; Nivolumab; Advanced Cancers; Small cell lung cancer; Squamous non-small cell lung cancer; LSD1 inhibitor
MeSH Terms: conditions — Neoplasms; Small Cell Lung Carcinoma | interventions — pulrodemstat besilate; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A: SCLC in ICI naïve subjects (Experimental): CC-90011 will be given orally (PO) at a dose of 40 mg on a once weekly basis in a continuous 28-day cycle.
  Nivolumab will be administered intravenously at a dose of 480 mg every 4 weeks per local practice as a 30 minute or a 60-minute infusion as per local practice.
  Interventions: Drug: CC-90011; Drug: Nivolumab
- Cohort B: SCLC in ICI progressor subjects (Experimental): CC-90011 will be given orally (PO) at a dose of 40 mg on a once weekly basis in a continuous 28-day cycle.
  Nivolumab will be administered intravenously at a dose of 480 mg every 4 weeks per local practice as a 30 minute or a 60-minute infusion as per local practice.
  Interventions: Drug: CC-90011; Drug: Nivolumab
- Cohort C: sqNSCLC in ICI progressor subjects (Experimental): CC-90011 will be given orally (PO) at a dose of 40 mg on a once weekly basis in a continuous 28-day cycle.
  Nivolumab will be administered intravenously at a dose of 480 mg every 4 weeks per local practice as a 30 minute or a 60-minute infusion as per local practice.
  Interventions: Drug: CC-90011; Drug: Nivolumab

INTERVENTIONS:
Drug: CC-90011 — CC-90011
Drug: Nivolumab — Nivolumab

SUMMARY:
This is a Phase 2, multicenter, open-label, multi-cohort study to assess safety and efficacy of CC-90011 in combination with nivolumab in subjects with small cell lung cancer or squamous non-small cell lung cancer who have progressed after 1 or 2 lines of therapies.

The primary objectives of the study are to evaluate the overall response rate of subjects treated with CC-90011 in combination with nivolumab in three cohorts:

* Cohort A: SCLC in ICI naïve subjects
* Cohort B: SCLC in ICI progressor subjects
* Cohort C: sqNSCLC in ICI progressor subjects Overall response rate is defined as the proportion of subjects in the treated population who had complete response (CR) or partial response (PR) as assessed by Investigator review per RECIST v1.1.

In Cohort A, expected ORR for nivolumab monotherapy is 14% while target ORR is 30%. To achieve at least 80% power with one-sided type 1 error 0.1, 39 subjects will be enrolled according to a 2-stage group sequential design based on a binomial test. In stage 1, 12 subjects will be enrolled and treated with CC-90011 in combination with nivolumab. If there are 2 or more subjects responding, Cohort A will continue to enroll an additional 27 subjects. If 1 or less subjects respond in stage 1, Cohort A will stop for futility.

In Cohort B and C, expected ORR for nivolumab monotherapy is 5% while target ORR is 15%. To achieve at least 80% power with one-sided type 1 error 0.1, 48 subjects will be enrolled according to a 2-stage group sequential design based on a binomial test. In stage 1, 14 subjects will be enrolled and treated with CC-90011 in combination with nivolumab. If there are 1 or more subjects responding, Cohort B and C will continue to enroll an additional 34 subjects each. If 0 subjects respond in stage 1, Cohort B and C will stop for futility.

ELIGIBILITY:
Inclusion Criteria:

Subjects must satisfy the following criteria to be enrolled in the study:

1. Subject is ≥ 18 years of age at the time of signing the informed consent form (ICF).
2. Subject with histological or cytological confirmation of extensive stage Small Cell Lung Cancer (ES SCLC) or Stage IIIb or IV squamous Non-Small Cell Lung Cancer (sqNSCLC)
3. Subject has received 1 or 2 prior lines of therapies, defined as:

   1. Cohort A (SCLC, Immune Checkpoint Inhibitor naïve):

      * At least 1 prior treatment including a platinum-based chemotherapy doublet
      * A minimum of 3 cycles of platinum-based chemotherapy in first line treatment, unless stopped at 2 cycles due to treatment-related toxicity
   2. Cohort B (SCLC, ICI progressors):

      * At least 1 prior first or second line treatment includes an ICI
      * If treatment includes an ICI as maintenance therapy, at least 1 cycle of ICI in maintenance should have been completed
      * At least 1 prior treatment including a platinum-based chemotherapy doublet
      * A minimum of 3 cycles of platinum-based chemotherapy, with or without ICI, in first line treatment, unless stopped at 2 cycles due to treatment-related toxicity
      * Subject must have progressed during ICI therapy, defined as unequivocal progression on or within 3 months of the last dose of ICI therapy (if no subsequent therapy)
   3. Cohort C (sqNSCLC, ICI progressors):

      * At least 1 prior first or second line treatment includes an ICI
      * If treatment includes an ICI as maintenance therapy, at least 1 cycle of ICI in maintenance should have been completed
      * At least 1 prior treatment including a platinum-based chemotherapy doublet
      * A minimum of 3 cycles of platinum-based chemotherapy, with or without an ICI, in first line treatment, unless stopped at 2 cycles due to treatment-related toxicity
      * Subject must have progressed during ICI therapy, defined as unequivocal progression on or within 3 months of the last dose of ICI therapy (if no subsequent therapy)
4. Subject has progressed at the last line of therapy.
5. Subject has a measurable disease defined by RECIST v1.1.
6. Subject agrees to provide a tumor biopsy from primary or metastatic site prior to first dose and at a pre-specified timepoint during treatment. Core biopsy is required however, in the event a core biopsy may not otherwise be feasible in the opinion of the treating physician, an endobronchial ultrasound-guided fine needle aspirate [EBUS-FNA]) biopsy, using the largest gauge needle, may be performed instead.
7. Subject has ECOG Performance Status of 0 to 1.
8. Subject must have the following laboratory values:

   1. Absolute neutrophil count (ANC) ≥ 1.5 x 109/L
   2. Hemoglobin (Hgb) ≥ 9 g/dL (one-time blood transfusion is allowed)
   3. Platelet (Plt) Count ≥ 150 x 109/L
   4. White blood cells (WBC) ≥ 2 x 109L
   5. Serum AST/serum glutamic oxaloacetic transaminase (SGOT) or ALT/serum glutamic pyruvic transaminase (SGPT) ≤ 3 x upper limit of normal (ULN) or ≤ 5 x ULN if presence of liver metastases
   6. Total serum bilirubin ≤ 1.5 x ULN (≤ 3 x ULN, if Gilbert's syndrome or if indirect bilirubin concentrations are suggestive of extrahepatic source of the elevation)
   7. Creatinine clearance (CrCl) ≥ 60 mL/minute based on Cockcroft-Gault or modification of diet in renal disease (MDRD) or ≥ 60 mL/min/1.73 m2

Exclusion Criteria:

The presence of any of the following will exclude a subject from enrollment:

1. Subject has not recovered to Grade 2 or lower clinically significant toxicities related to the prior therapy (alopecia excluded).
2. Subject has received prior LSD1 therapies.
3. Subject has a history of severe hypersensitivity reactions to other monoclonal antibodies
4. Subject with symptomatic and untreated or unstable central nervous system (CNS) metastases.

   1. Subject has recently been treated with whole brain radiation or stereotactic radiosurgery for CNS metastases must have completed therapy at least 2 weeks prior to Cycle 1 Day 1 and has a follow-up brain computed tomography (CT) or magnetic resonance imaging (MRI) demonstrating either stable or improving metastases 2 or more weeks after completion of radiotherapy.
   2. Subject must be asymptomatic and off steroids or on stable dose of steroids for at least 2 weeks (≤ 10 mg daily prednisone or equivalent) prior to first dose.
5. Subject has persistent diarrhea due to a malabsorptive syndrome (such as celiac sprue or inflammatory bowel disease) ≥ NCI CTCAE Grade 2, despite medical management), or any other significant gastrointestinal (GI) disorder that could affect the absorption of the study treatments.
6. Subject with symptomatic or uncontrolled ulcers (gastric or duodenal), particularly those with a history of and/or risk of perforation and GI tract hemorrhages.
7. Subject with any hemorrhage/bleeding event > NCI CTCAE Grade 2 or haemoptysis > 1 teaspoon within 4 weeks prior to the first dose.
8. Subject has any of the following cardiovascular criteria:

   1. Evidence of acute or ongoing cardiac ischemia
   2. Current symptomatic pulmonary embolism
   3. Unstable angina pectoris or myocardial infarction ≤ 6 months prior to enrollment
   4. Heart failure of New York Heart Association Classification III or IV ≤ 6 months prior to enrollment
   5. Persistent or clinically meaningful ventricular arrhythmias prior to enrollment
   6. Cerebral vascular accident or transient ischemic attack ≤ 6 months prior to enrollment
   7. QT corrected based on Fridericia's equation (QTcF) ≥ 450 milliseconds (msec) on Screening ECG, a baseline prolongation of QTcF interval ≥ 450 msec (NCI CTCAE Grade ≥ 2)
   8. A history of additional risk factors for Torsades de pointes (TdP) (eg, heart failure, hypokalemia, family history of Long QT Syndrome)
   9. Uncontrolled hypertension (blood pressure ≥ 160/95 mm Hg)
9. Subject has known human immunodeficiency virus (HIV) infection.
10. Subject has known chronic active hepatitis B or C virus (HBV, HCV) infection.

    1. Subject who is seropositive due to HBV vaccination is eligible.
    2. Subject who has no active viral infection and is under adequate prophylaxis against HBV reactivation is eligible.
11. Subject has any other malignancy within 2 years prior to enrollment, with the exception of adequately treated in-situ bladder cancer, in-situ carcinoma of the cervix, uteri, nonmelanomatous skin cancer, ductal in situ breast carcinoma, thyroid cancer, or early stage prostate cancer (all treatment of which should have been completed 6 months prior to enrollment).
12. Subject has medical conditions requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone or equivalent) or other immunosuppressive medications within 14 days of enrollment.

    1. A brief (≤ 7 days) course of corticosteroids for prophylaxis (eg, contrast dye allergy) or for treatment of nonautoimmune conditions (eg, delayed-type hypersensitivity reaction caused by contact allergen) is permitted.
    2. Adrenal replacement steroid doses > 10 mg daily prednisone or equivalent are permitted in the absence of active autoimmune disease.
    3. Topical, ocular, intra-articular, intranasal, and inhalational corticosteroids (with minimal systemic absorption) are permitted.
13. Subject has active autoimmune diseases or history of autoimmune diseases that may relapse. Subjects with the following diseases are allowed to be enrolled after further screening: type I diabetes, hypothyroidism managed with hormone replacement therapy only, skin diseases not requiring systemic treatment (such as vitiligo, psoriasis, or alopecia), or diseases not expected to recur in the absence of external triggering factors.
14. Subject is pregnant or nursing.
15. Subject has a history of persistent skin rash ≥ NCI CTCAE Grade 2 related to prior ICI therapy.
16. Subject has organ transplant history, including allogeneic stem cell transplant.
17. Subject has interstitial lung disease history.
18. Subject has received a live/attenuated vaccine within 30 days of first dose.
19. Subject has previous SARS-CoV-2 infection either suspected or confirmed within 4 weeks prior to screening.

    1. Acute symptoms must have resolved and based on Investigator assessment in consultation with the Medical Monitor, there are no sequelae that would place the subject at a higher risk of receiving investigational treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2020-07-14 (Actual); Primary Completion 2023-12-19 (Actual); Study Completion 2023-12-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (37):
- United States (8):
  - Local Institution - 102, Indianapolis, Indiana
  - Local Institution - 106, New York, New York
  - Local Institution - 105, Canton, Ohio
  - Local Institution - 104, Cleveland, Ohio
  - Local Institution - 109, Pittsburgh, Pennsylvania
  - Local Institution - 107, Fort Sam Houston, Texas
  - Local Institution - 110, Houston, Texas
  - Local Institution - 111, Fairfax, Virginia
- France (5):
  - Local Institution - 156, Lyon
  - Local Institution - 153, Marseille
  - Local Institution - 154, Rennes
  - Local Institution - 151, Saint-Herblain
  - Local Institution - 152, Villejuif
- Italy (5):
  - Local Institution - 301, Aviano
  - Local Institution - 306, Meldola
  - Local Institution - 303, Milan
  - Local Institution - 305, Roma
  - Local Institution - 304, Verona
- Poland (4):
  - Local Institution - 451, Lodz
  - Local Institution - 452, Lodz
  - Local Institution - 454, Poznan
  - Local Institution - 453, Warsaw
- Spain (12):
  - Local Institution - 361, A Coruña
  - Local Institution - 351, Badalona (Barcelona)
  - Local Institution - 355, Barcelona
  - Local Institution - 356, Barcelona
  - Local Institution - 359, Las Palmas de Gran Canaria
  - Local Institution - 358, Madrid
  - Local Institution - 353, Madrid
  - Local Institution - 357, Madrid
  - Local Institution - 360, Majadahonda, Madrid
  - Local Institution - 352, Pamplona
  - Local Institution - 362, Valencia
  - Local Institution - 354, Valencia
- United Kingdom (3):
  - Local Institution - 254, London
  - Local Institution - 251, Manchester
  - Local Institution - 255, Sutton-Surrey

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — http://www.BMSStudyConnect.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort A 40 mg: Participants with small cell lung cancer (SCLC) and immune checkpoint inhibitor (ICI) naive received capsule of 40 milligram (mg) of CC-90011 orally once in a week in a continuous 28-day cycle. Nivolumab were administered intravenously at a dose of 480 mg every 4 weeks as a 30 minute or a 60-minute intravenous infusion.
- Cohort A 60mg: Participants with SCLC and ICI naive received capsule of 60 mg of CC-90011 orally once in a week in a continuous 28-day cycle. Nivolumab were administered intravenously at a dose of 480 mg every 4 weeks as a 30 minute or a 60-minute intravenous infusion.
- Cohort B 40 mg: Participants with SCLC and ICI progressor received capsule of 40 mg of CC-90011 orally once in a week in a continuous 28-day cycle. Nivolumab were administered intravenously at a dose of 480 mg every 4 weeks as a 30 minute or a 60-minute intravenous infusion.
- Cohort C: Participants with squamous non-small cell lung cancer (sqNSCLC) and ICI progressor received capsule of 40 mg of CC-90011 orally once in a week in a continuous 28-day cycle. Nivolumab were administered intravenously at a dose of 480 mg every 4 weeks as a 30 minute or a 60-minute intravenous infusion.
Period: Overall Study
Arm/Group | Cohort A 40 mg | Cohort A 60mg | Cohort B 40 mg | Cohort C
Started | 39 | 2 | 14 | 37
Completed | 8 | 0 | 0 | 2
Not Completed | 31 | 2 | 14 | 35
Not completed — Other reason | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 2
Not completed — Withdrawal by Subject | 4 | 0 | 1 | 4
Not completed — Adverse Event | 0 | 0 | 0 | 2
Not completed — Death | 27 | 2 | 13 | 26

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A 40 mg | Cohort A 60mg | Cohort B 40 mg | Cohort C | Total
Number analyzed (Participants) | 39 | 2 | 14 | 37 | 92
Age, Customized [Number; unit: participants]
  < 65 years | 21 | 2 | 11 | 17 | 51
  >= 65 - < 75 years | 16 | 0 | 3 | 15 | 34
  >= 75 years | 2 | 0 | 0 | 5 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 0 | 5 | 2 | 18
  Male | 28 | 2 | 9 | 35 | 74
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2 | 3 | 7
  Not Hispanic or Latino | 30 | 2 | 7 | 23 | 62
  Unknown or Not Reported | 7 | 0 | 5 | 11 | 23
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 33 | 2 | 9 | 28 | 72
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 6 | 0 | 5 | 9 | 20

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: Overall response rate was defined as the percentage of participants in the treated population who had confirmed complete response (CR) or confirmed partial response (PR) as assessed by Investigator review per RECIST v1.1. CR was defined as disappearance of all target lesions and any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 millimeter (mm). PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. Disease progression (PD) is defined as an additional 10% increase in tumor burden with a minimum 5 mm absolute increase from time of initial PD. This includes an increase in the sum of diameters of all target lesions and/or the diameters of new measurable lesions compared to the time of the initial PD.
Time Frame: Every 6 weeks post Cycle 1 (each cycle is of 28 days) Day 1 for the first 24 weeks and then every 8 weeks until disease progression, new anticancer therapy, death or withdrawal by participants (up to approximately 33 months)
Population: Treated population consist of all participants who enrolled and took at least one dose of either CC-90011 or nivolumab.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort A 40 mg | Cohort A 60mg | Cohort B 40 mg | Cohort C
Number analyzed (Participants) | 39 | 2 | 14 | 35
percentage of participants | 10.3 [2.9 to 24.2] | 0 [0.0 to 84.2] | 0 [0.0 to 23.2] | 8.6 [1.8 to 23.1]

2. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events by Maximal National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE)
Description: An Adverse Event (AE) is defined as any new untoward medical occurrence or worsening of a preexisting medical condition in a clinical investigation participant administered study treatment and that does not necessarily have a causal relationship with this treatment. Treatment-emergent Adverse Events are defined as any AEs that begin or worsen on or after the start of study drug through 28 days after the last dose of CC-90011 or until 100 days after last dose of nivolumab study treatment. AEs were graded using the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 (Grade 1=mild, Grade 2=Moderate, Grade 3 = Severe, Grade 4 = Life-threatening, Grade 5 = Death).
Time Frame: From the start of study drug through 28 days after the last dose of CC-90011 or until 100 days after last dose of Nivolumab (up to 849 days)
Population: Treated population consist of all participants who enrolled and took at least one dose of either CC-90011 or nivolumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A 40 mg | Cohort A 60mg | Cohort B 40 mg | Cohort C
Number analyzed (Participants) | 39 | 2 | 14 | 35
Participants
  Grade 1 | 0 | 0 | 2 | 1
  Grade 2 | 14 | 0 | 2 | 4
  Grade 3 | 7 | 0 | 3 | 20
  Grade 4 | 8 | 2 | 2 | 3
  Grade 5 | 10 | 0 | 5 | 6
  Missing | 0 | 0 | 0 | 1

3. Secondary Outcome: Number of Participants With Laboratory Results With CTCAE Toxicity Grade >=3 for Hematology Parameters
Description: Laboratory results were graded using the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 (Grade 3 =Severe, Grade 4 = Life-threatening).
Time Frame: Cycle 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 14 and 18 (each cycle is of 28 days)
Population: Treated population consist of all participants who enrolled and took at least one dose of either CC-90011 or nivolumab
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A 40 mg | Cohort A 60mg | Cohort B 40 mg | Cohort C
Number analyzed (Participants) | 39 | 2 | 14 | 35
Participants
  Cycle 1 Hemoglobin | 3 | 0 | 1 | 3
  Cycle 1 Leukocytes | 1 | 0 | 0 | 0
  Cycle 1 Lymphocytes | 5 | 0 | 3 | 3
  Cycle 1 Neutrophils | 1 | 1 | 0 | 0
  Cycle 1 Platelets | 3 | 2 | 1 | 0
  Cycle 2 Hemoglobin | 1 | 0 | 0 | 1
  Cycle 2 Lymphocytes | 3 | 0 | 0 | 2
  Cycle 2 Platelets | 5 | 0 | 0 | 1
  Cycle 3 Lymphocytes | 1 | 0 | 1 | 3
  Cycle 3 Platelets | 1 | 0 | 0 | 0
  Cycle 4 Lymphocytes | 1 | 0 | 0 | 1
  Cycle 5 Hemoglobin | 1 | 0 | 0 | 0
  Cycle 5 Lymphocytes | 2 | 0 | 0 | 1
  Cycle 6 Lymphocytes | 1 | 0 | 0 | 1
  Cycle 6 Platelets | 1 | 0 | 0 | 0
  Cycle 7 Lymphocytes | 0 | 0 | 0 | 1
  Cycle 8 Lymphocytes | 0 | 0 | 0 | 1
  Cycle 8 Platelets | 1 | 0 | 0 | 0
  Cycle 9 Lymphocytes | 0 | 0 | 0 | 1
  Cycle 9 Platelets | 1 | 0 | 0 | 0
  Cycle 10 Lymphocytes | 0 | 0 | 0 | 1
  Cycle 10 Platelets | 1 | 0 | 0 | 0
  Cycle 11 Lymphocytes | 0 | 0 | 0 | 1
  Cycle 12 Hemoglobin | 1 | 0 | 0 | 0
  Cycle 14 Platelets | 1 | 0 | 0 | 0
  Cycle 18 Neutrophils | 0 | 0 | 0 | 1
  Cycle 18 Platelets | 0 | 0 | 0 | 1

4. Secondary Outcome: Number of Participants With Laboratory Results With CTCAE Toxicity Grade >=3 for Chemistry Parameters
Description: as for outcome 3
Time Frame: Cycle 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 14 and 18 (Each cycle is of 28 days)
Population: Treated population consist of all participants who enrolled and took at least one dose of either CC-90011 or nivolumab
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A 40 mg | Cohort A 60mg | Cohort B 40 mg | Cohort C
Number analyzed (Participants) | 39 | 2 | 14 | 35
Participants
  Cycle 1 Alanine Aminotransferase | 0 | 0 | 2 | 0
  Cycle 1 Albumin | 0 | 0 | 0 | 1
  Cycle 1 Alkaline Phosphatase | 0 | 0 | 0 | 1
  Cycle 1 Aspartate Aminotransferase | 0 | 0 | 1 | 1
  Cycle 1 Bilirubin | 1 | 0 | 0 | 1
  Cycle 1 Direct Bilirubin | 1 | 0 | 2 | 1
  Cycle 1 Sodium | 3 | 1 | 1 | 1
  Cycle 2 Alanine Aminotransferase | 1 | 0 | 1 | 0
  Cycle 2 Alkaline Phosphatase | 0 | 0 | 1 | 0
  Cycle 2 Aspartate Aminotransferase | 1 | 0 | 1 | 0
  Cycle 2 Direct Bilirubin | 1 | 0 | 1 | 0
  Cycle 2 Glucose | 0 | 0 | 0 | 1
  Cycle 2 Sodium | 1 | 1 | 0 | 1
  Cycle 3 Calcium | 0 | 0 | 0 | 1
  Cycle 3 Direct Bilirubin | 0 | 0 | 1 | 0
  Cycle 3 Glucose | 0 | 0 | 0 | 1
  Cycle 3 Potassium | 0 | 0 | 1 | 0
  Cycle 4 Direct Bilirubin | 0 | 0 | 1 | 0
  Cycle 4 Sodium | 1 | 0 | 0 | 0
  Cycle 5 Direct Bilirubin | 0 | 0 | 1 | 0
  Cycle 6 Calcium | 1 | 0 | 0 | 0
  Cycle 6 Direct Bilirubin | 0 | 0 | 1 | 0
  Cycle 6 Sodium | 0 | 0 | 0 | 1
  Cycle 7 Direct Bilirubin | 0 | 0 | 1 | 0
  Cycle 8 Direct Bilirubin | 0 | 0 | 1 | 0
  Cycle 9 Direct Bilirubin | 0 | 0 | 1 | 0
  Cycle 9 Glucose | 0 | 0 | 0 | 1
  Cycle 10 Direct Bilirubin | 0 | 0 | 1 | 0
  Cycle 11 Direct Bilirubin | 0 | 0 | 1 | 0
  Cycle 14 Direct Bilirubin | 1 | 0 | 0 | 0
  Cycle 14 Sodium | 1 | 0 | 0 | 0
  Cycle 16 Potassium | 1 | 0 | 0 | 0

5. Secondary Outcome: Number of Participants Receiving Concomitant Medication
Description: Concomitant medication is defined as medications that were either initiated before the first dose of study drug and continued during the study treatment, or initiated on/after the date of the first dose of study drug and on/before the date of treatment discontinuation.
Time Frame: From first dose till treatment discontinuation due to any reason (Up to approximately 107 weeks)
Population: Treated population consist of all participants who enrolled and took at least one dose of either CC-90011 or nivolumab
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A 40 mg | Cohort A 60mg | Cohort B 40 mg | Cohort C
Number analyzed (Participants) | 39 | 2 | 14 | 35
Participants | 39 | 2 | 14 | 35

6. Secondary Outcome: Change From Baseline at End of Treatment in Vital Sign - Weight
Description: Baseline value was defined as the last non-missing value on or before the day that first dose of study drug is administered; if multiple values are present for the same date, the average of these values will be used as the baseline.
Time Frame: Baseline and End of Treatment (Up to 107 weeks)
Population: Treated population consist of all participants who enroll and take at least one dose of either CC-90011 or nivolumab. Participants with weight measurements available at the specific timepoint were analyzed.
Measure: Mean (Standard Deviation); unit: kilogram
Arm/Group | Cohort A 40 mg | Cohort A 60mg | Cohort B 40 mg | Cohort C
Number analyzed (Participants) | 32 | 1 | 10 | 21
kilogram | -1.88 (5.583) | -1.00 (NA) — Standard Deviation is not available as only 1 participant was analyzed. | -2.58 (5.651) | -4.20 (8.065)

7. Secondary Outcome: Change From Baseline at End of Treatment in Vital Sign - Diastolic Blood Pressure (DBP) and Systolic Blood Pressure (SBP)
Description: as for outcome 6
Time Frame: Baseline and End of Treatment (Up to 107 weeks)
Population: Treated population consist of all participants who enrolled and took at least one dose of either CC-90011 or nivolumab. Participants with DBP and SBP measurements available at the specific timepoint were analyzed.
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Arm/Group | Cohort A 40 mg | Cohort A 60mg | Cohort B 40 mg | Cohort C
Number analyzed (Participants) | 31 | 1 | 11 | 24
millimeters of mercury (mmHg)
  Systolic Blood Pressure | -8.5 (18.35) | 5.0 (NA) — Standard Deviation is not available as only 1 participant was analyzed. | 4.8 (14.82) | -11.2 (15.19)
  Diastolic Blood Pressure | -4.9 (10.84) | 9.0 (NA) — Standard Deviation is not available as only 1 participant was analyzed. | -3.2 (6.60) | -3.1 (9.89)

8. Secondary Outcome: Change From Baseline at End of Treatment in Vital Sign - Temperature
Description: as for outcome 6
Time Frame: Baseline and End of Treatment (Up to 107 weeks)
Population: Treated population consist of all participants who enrolled and took at least one dose of either CC-90011 or nivolumab. Participants with temperature measurements available at the specific timepoint were analyzed.
Measure: Mean (Standard Deviation); unit: degree Celsius
Arm/Group | Cohort A 40 mg | Cohort A 60mg | Cohort B 40 mg | Cohort C
Number analyzed (Participants) | 31 | 1 | 11 | 23
degree Celsius | 0.01 (0.376) | 0.20 (NA) — Standard Deviation is not available as only 1 participant was analyzed. | 0.03 (0.388) | -0.04 (0.509)

9. Secondary Outcome: Change From Baseline at End of Treatment in Vital Sign - Pulse Rate
Description: as for outcome 6
Time Frame: Baseline and End of Treatment (Up to 107 weeks)
Population: Treated population consist of all participants who enrolled and took at least one dose of either CC-90011 or nivolumab. Participants with pulse rate measurements available at the specific timepoint were analyzed.
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Cohort A 40 mg | Cohort A 60mg | Cohort B 40 mg | Cohort C
Number analyzed (Participants) | 31 | 1 | 10 | 24
beats per minute | -1.0 (12.37) | -8.0 (NA) — Standard Deviation is not available as only 1 participant was analyzed. | 12.0 (14.73) | 0.4 (16.58)

10. Secondary Outcome: Number of Participants With Post-Baseline Grade Shift in Eastern Cooperative Oncology Group Performance (ECOG) Status
Description: ECOG Scale was used to assess performance status. Grades: 0: Fully active, able to carry on all pre-disease performance without restriction. 1: Restricted in physically strenuous activity but ambulatory, able to carry out work of light nature. 2: Ambulatory, capable of self-care, unable to carry out work activities. Up and about more than 50% waking hours. 3: Capable of limited self-care, confined to bed/chair more than 50% waking hours. 4: Completely disabled. Cannot carry on any self-care. Totally confined to bed/chair. 5: Dead. Baseline value was defined as the last non-missing value on or before the day that first dose of study drug is administered; if multiple values are present for the same date, the average of these values will be used as the baseline.
Time Frame: Baseline and up to End of Treatment (107 weeks)
Population: Treated population consist of all participants who enrolled and took at least one dose of either CC-90011 or nivolumab. Participants with ECOG measurements available at the specific timepoint were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A 40 mg | Cohort A 60mg | Cohort B 40 mg | Cohort C
Number analyzed (Participants) | 33 | 1 | 11 | 23
Participants
  Grade 0 to Grade 0: number analyzed (Participants) | 9 | 0 | 5 | 7
  Grade 0 to Grade 0 | 2 | 0 | 4 | 1
  Grade 0 to Grade 1: number analyzed (Participants) | 9 | 0 | 5 | 7
  Grade 0 to Grade 1 | 6 | 0 | 1 | 3
  Grade 0 to Grade 2: number analyzed (Participants) | 9 | 0 | 5 | 7
  Grade 0 to Grade 2 | 1 | 0 | 0 | 2
  Grade 0 to Grade 3: number analyzed (Participants) | 9 | 0 | 5 | 7
  Grade 0 to Grade 3 | 0 | 0 | 0 | 1
  Grade 0 to Grade 4: number analyzed (Participants) | 9 | 0 | 5 | 7
  Grade 0 to Grade 4 | 0 | 0 | 0 | 0
  Grade 0 to Grade 5: number analyzed (Participants) | 9 | 0 | 5 | 7
  Grade 0 to Grade 5 | 0 | 0 | 0 | 0
  Grade 1 to Grade 0: number analyzed (Participants) | 24 | 1 | 6 | 16
  Grade 1 to Grade 0 | 0 | 0 | 0 | 0
  Grade 1 to Grade 1: number analyzed (Participants) | 24 | 1 | 6 | 16
  Grade 1 to Grade 1 | 17 | 1 | 5 | 8
  Grade 1 to Grade 2: number analyzed (Participants) | 24 | 1 | 6 | 16
  Grade 1 to Grade 2 | 7 | 0 | 0 | 5
  Grade 1 to Grade 3: number analyzed (Participants) | 24 | 1 | 6 | 16
  Grade 1 to Grade 3 | 0 | 0 | 1 | 3
  Grade 1 to Grade 4: number analyzed (Participants) | 24 | 1 | 6 | 16
  Grade 1 to Grade 4 | 0 | 0 | 0 | 0
  Grade 1 to Grade 5: number analyzed (Participants) | 24 | 1 | 6 | 16
  Grade 1 to Grade 5 | 0 | 0 | 0 | 0
  Grade 2 to Grade 0: number analyzed (Participants) | 0 | 0 | 0 | 0
  Grade 2 to Grade 0 | 0 | 0 | 0 | 0
  Grade 2 to Grade 1: number analyzed (Participants) | 0 | 0 | 0 | 0
  Grade 2 to Grade 1 | 0 | 0 | 0 | 0
  Grade 2 to Grade 2: number analyzed (Participants) | 0 | 0 | 0 | 0
  Grade 2 to Grade 2 | 0 | 0 | 0 | 0
  Grade 2 to Grade 3: number analyzed (Participants) | 0 | 0 | 0 | 0
  Grade 2 to Grade 3 | 0 | 0 | 0 | 0
  Grade 2 to Grade 4: number analyzed (Participants) | 0 | 0 | 0 | 0
  Grade 2 to Grade 4 | 0 | 0 | 0 | 0
  Grade 2 to Grade 5: number analyzed (Participants) | 0 | 0 | 0 | 0
  Grade 2 to Grade 5 | 0 | 0 | 0 | 0
  Grade 3 to Grade 0: number analyzed (Participants) | 0 | 0 | 0 | 0
  Grade 3 to Grade 0 | 0 | 0 | 0 | 0
  Grade 3 to Grade 1: number analyzed (Participants) | 0 | 0 | 0 | 0
  Grade 3 to Grade 1 | 0 | 0 | 0 | 0
  Grade 3 to Grade 2: number analyzed (Participants) | 0 | 0 | 0 | 0
  Grade 3 to Grade 2 | 0 | 0 | 0 | 0
  Grade 3 to Grade 3: number analyzed (Participants) | 0 | 0 | 0 | 0
  Grade 3 to Grade 3 | 0 | 0 | 0 | 0
  Grade 3 to Grade 4: number analyzed (Participants) | 0 | 0 | 0 | 0
  Grade 3 to Grade 4 | 0 | 0 | 0 | 0
  Grade 3 to Grade 5: number analyzed (Participants) | 0 | 0 | 0 | 0
  Grade 3 to Grade 5 | 0 | 0 | 0 | 0
  Grade 4 to Grade 0: number analyzed (Participants) | 0 | 0 | 0 | 0
  Grade 4 to Grade 0 | 0 | 0 | 0 | 0
  Grade 4 to Grade 1: number analyzed (Participants) | 0 | 0 | 0 | 0
  Grade 4 to Grade 1 | 0 | 0 | 0 | 0
  Grade 4 to Grade 2: number analyzed (Participants) | 0 | 0 | 0 | 0
  Grade 4 to Grade 2 | 0 | 0 | 0 | 0
  Grade 4 to Grade 3: number analyzed (Participants) | 0 | 0 | 0 | 0
  Grade 4 to Grade 3 | 0 | 0 | 0 | 0
  Grade 4 to Grade 4: number analyzed (Participants) | 0 | 0 | 0 | 0
  Grade 4 to Grade 4 | 0 | 0 | 0 | 0
  Grade 4 to Grade 5: number analyzed (Participants) | 0 | 0 | 0 | 0
  Grade 4 to Grade 5 | 0 | 0 | 0 | 0
  Grade 5 to Grade 0: number analyzed (Participants) | 0 | 0 | 0 | 0
  Grade 5 to Grade 0 | 0 | 0 | 0 | 0
  Grade 5 to Grade 1: number analyzed (Participants) | 0 | 0 | 0 | 0
  Grade 5 to Grade 1 | 0 | 0 | 0 | 0
  Grade 5 to Grade 2: number analyzed (Participants) | 0 | 0 | 0 | 0
  Grade 5 to Grade 2 | 0 | 0 | 0 | 0
  Grade 5 to Grade 3: number analyzed (Participants) | 0 | 0 | 0 | 0
  Grade 5 to Grade 3 | 0 | 0 | 0 | 0
  Grade 5 to Grade 4: number analyzed (Participants) | 0 | 0 | 0 | 0
  Grade 5 to Grade 4 | 0 | 0 | 0 | 0
  Grade 5 to Grade 5: number analyzed (Participants) | 0 | 0 | 0 | 0
  Grade 5 to Grade 5 | 0 | 0 | 0 | 0

11. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events Leading to Dose Reduction of CC-90011
Description: Adverse Event (AE) is defined as any new untoward medical occurrence or worsening of a preexisting medical condition in a clinical investigation participant administered study treatment and that does not necessarily have a causal relationship with this treatment. Treatment-emergent Adverse Events are defined as any AEs that begin or worsen on or after the start of study drug through 28 days after the last dose of CC-90011 or until 100 days after last dose of nivolumab study treatment.
Time Frame: as for outcome 2
Population: Treated population consist of all participants who enrolled and took at least one dose of either CC-90011 or nivolumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A 40 mg | Cohort A 60mg | Cohort B 40 mg | Cohort C
Number analyzed (Participants) | 39 | 2 | 14 | 35
Participants | 7 | 2 | 3 | 6

12. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events Leading to Dose Interruption of CC-90011
Description: as for outcome 11
Time Frame: as for outcome 2
Population: Treated population consist of all participants who enrolled and took at least one dose of either CC-90011 or nivolumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A 40 mg | Cohort A 60mg | Cohort B 40 mg | Cohort C
Number analyzed (Participants) | 39 | 2 | 14 | 35
Participants | 27 | 1 | 6 | 26

13. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events Leading to Dose Interruption of Nivolumab
Description: as for outcome 11
Time Frame: From the start of study drug until 100 days after last dose of Nivolumab (up to 849 days)
Population: Treated population consist of all participants who enrolled and took at least one dose of either CC-90011 or nivolumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A 40 mg | Cohort A 60mg | Cohort B 40 mg | Cohort C
Number analyzed (Participants) | 39 | 2 | 14 | 35
Participants | 16 | 0 | 3 | 14

14. Secondary Outcome: Duration of Response
Description: Duration of Response was defined as the time from the first occurrence of a confirmed documented response to the time of the first documented tumor progression, as determined by Investigator review per RECIST v1.1, or death from any cause, whichever comes first. CR was defined as disappearance of all target lesions and any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 millimeter (mm). PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. Disease progression (PD) is defined as an additional 10% increase in tumor burden with a minimum 5 mm absolute increase from time of initial PD. This includes an increase in the sum of diameters of all target lesions and/or the diameters of new measurable lesions compared to the time of the initial PD.
Time Frame: Every 6 weeks post cycle 1 day 1 (each cycle is of 28 days) for the first 24 weeks and then every 8 weeks until disease progression, new anticancer therapy, death or withdrawal by participant (up to approximately 33 months))
Population: Treated population consist of all participants who enrolled and took at least one dose of either CC-90011 or nivolumab. Treated Population with confirmed Best Response of CR or PR were included in analysis.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Cohort A 40 mg | Cohort A 60mg | Cohort B 40 mg | Cohort C
Number analyzed (Participants) | 4 | 0 | 0 | 3
days | 645.0 (387.05) |  |  | 326.0 (201.14)

15. Secondary Outcome: Time to Response
Description: Time to response was defined as the time from the first dose of the study drug to the date of the first confirmed documented response (CR or PR), as assessed by Investigator review per RECIST v1.1. CR was defined as disappearance of all target lesions and any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 millimeter (mm). PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. Disease progression (PD) is defined as an additional 10% increase in tumor burden with a minimum 5 mm absolute increase from time of initial PD. This includes an increase in the sum of diameters of all target lesions and/or the diameters of new measurable lesions compared to the time of the initial PD.
Time Frame: as for outcome 14
Population: Treated population consist of all participants who enrolled and took at least one dose of either CC-90011 or nivolumab. Treated Population with confirmed best response of CR or PR.
Measure: Median (Full Range); unit: days
Arm/Group | Cohort A 40 mg | Cohort A 60mg | Cohort B 40 mg | Cohort C
Number analyzed (Participants) | 4 | 0 | 0 | 3
days | 82.0 [38 to 91] |  |  | 79.0 [38 to 126]

16. Secondary Outcome: Progression-Free Survival
Description: Progression-Free Survival is the time from first dose of study treatment to the date of the first objectively documented tumor progression as assessed by Investigator review per RECIST v1.1 or death from any cause, whichever occurs first. Disease progression (PD) is defined as an additional 10% increase in tumor burden with a minimum 5 mm absolute increase from time of initial PD. This includes an increase in the sum of diameters of all target lesions and/or the diameters of new measurable lesions compared to the time of the initial PD.
Time Frame: as for outcome 14
Population: Treated population consist of all participants who enrolled and took at least one dose of either CC-90011 or nivolumab.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Cohort A 40 mg | Cohort A 60mg | Cohort B 40 mg | Cohort C
Number analyzed (Participants) | 39 | 2 | 14 | 35
days | 126.4 (190.29) | 33.5 (7.78) | 65.6 (57.23) | 184.9 (202.20)

17. Secondary Outcome: Time to First Subsequent Therapy
Description: Time to First Subsequent Therapy was defined as the time from the first dose of the study drug to the date of the next cancer therapy or death.
Time Frame: From the first dose of study drug to the date of next cancer therapy or death due to any cause (up to approximately 33 months)
Population: Treated population consist of all participants who enrolled and took at least one dose of either CC-90011 or nivolumab.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Cohort A 40 mg | Cohort A 60mg | Cohort B 40 mg | Cohort C
Number analyzed (Participants) | 39 | 2 | 14 | 35
days | 181.3 (183.87) | 60.0 (2.83) | 113.3 (111.51) | 224.1 (203.26)

ADVERSE EVENTS:
Time Frame: All cause mortality was collected from first dose till death due to any cause (Up to approximately 33 months). Serious and Non-serious adverse events were collected from from the start of study drug through 28 days after the last dose of CC-90011 or until 100 days after last dose of Nivolumab (up to 849 days).
Description: All cause mortality was collected for all the enrolled participants. Serious and Non-Serious Adverse Events were collected for all the treated participants.
Arm/Group | Cohort A 40 mg | Cohort A 60mg | Cohort B 40 mg | Cohort C
All-Cause Mortality (participants affected / at risk) | 29/39 | 2/2 | 13/14 | 32/37
Serious Adverse Events (participants affected / at risk) | 20/39 | 2/2 | 8/14 | 25/35
Other Adverse Events (participants affected / at risk) | 39/39 | 2/2 | 14/14 | 33/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A 40 mg (N=39) | Cohort A 60mg (N=2) | Cohort B 40 mg (N=14) | Cohort C (N=35)
Anaemia (Blood and lymphatic system disorders) | 2 | 0 | 0 | 1
Haemolytic anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 2 | 0 | 0
Cardiac tamponade (Cardiac disorders) | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Gastric haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Umbilical hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Asthenia (General disorders) | 0 | 0 | 0 | 2
Chest pain (General disorders) | 0 | 0 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 0 | 1
General physical health deterioration (General disorders) | 5 | 0 | 4 | 3
Malaise (General disorders) | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 1 | 2
Hepatic failure (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Hepatitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 2
COVID-19 pneumonia (Infections and infestations) | 0 | 0 | 0 | 1
Empyema (Infections and infestations) | 1 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0 | 1 | 4
Respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0 | 0
General physical condition abnormal (Investigations) | 0 | 0 | 0 | 2
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 3 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Cervical cord compression (Nervous system disorders) | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 1 | 0
Bipolar disorder (Psychiatric disorders) | 1 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 1 | 0
Immune-mediated nephritis (Renal and urinary disorders) | 0 | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 3
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Hypovolaemic shock (Vascular disorders) | 1 | 0 | 0 | 0
Superior vena cava syndrome (Vascular disorders) | 0 | 0 | 0 | 1
Vena cava thrombosis (Vascular disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A 40 mg (N=39) | Cohort A 60mg (N=2) | Cohort B 40 mg (N=14) | Cohort C (N=35)
Anaemia (Blood and lymphatic system disorders) | 21 | 1 | 8 | 16
Leukopenia (Blood and lymphatic system disorders) | 2 | 0 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 5 | 0 | 0 | 4
Neutropenia (Blood and lymphatic system disorders) | 10 | 1 | 2 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 25 | 1 | 5 | 13
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 2
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 2
Hyperthyroidism (Endocrine disorders) | 3 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 6 | 0 | 0 | 0
Eyelid oedema (Eye disorders) | 0 | 0 | 1 | 0
Vision blurred (Eye disorders) | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 6 | 0 | 1 | 4
Abdominal pain upper (Gastrointestinal disorders) | 3 | 0 | 0 | 2
Constipation (Gastrointestinal disorders) | 6 | 0 | 2 | 5
Diarrhoea (Gastrointestinal disorders) | 8 | 0 | 0 | 5
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Dysphagia (Gastrointestinal disorders) | 2 | 0 | 0 | 2
Haematochezia (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 3 | 0 | 2 | 3
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 2 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 2 | 0 | 2 | 5
Asthenia (General disorders) | 9 | 0 | 5 | 12
Chest discomfort (General disorders) | 0 | 0 | 1 | 0
Chest pain (General disorders) | 0 | 1 | 0 | 0
Device related thrombosis (General disorders) | 0 | 0 | 1 | 0
Fatigue (General disorders) | 16 | 1 | 1 | 4
Gait disturbance (General disorders) | 2 | 0 | 0 | 1
Generalised oedema (General disorders) | 0 | 0 | 1 | 0
Mucosal inflammation (General disorders) | 1 | 0 | 0 | 2
Oedema peripheral (General disorders) | 4 | 0 | 1 | 0
Pyrexia (General disorders) | 1 | 0 | 4 | 9
Swelling (General disorders) | 0 | 0 | 1 | 1
Unevaluable event (General disorders) | 0 | 1 | 0 | 0
Hepatic cytolysis (Hepatobiliary disorders) | 0 | 0 | 2 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 3 | 0 | 0 | 1
Contrast media reaction (Immune system disorders) | 0 | 0 | 1 | 0
COVID-19 (Infections and infestations) | 3 | 0 | 0 | 6
Folliculitis (Infections and infestations) | 0 | 0 | 1 | 0
Implant site infection (Infections and infestations) | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 2 | 3
Respiratory tract infection (Infections and infestations) | 2 | 0 | 0 | 1
Tooth abscess (Infections and infestations) | 0 | 0 | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 3 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 7 | 1 | 2 | 3
Aspartate aminotransferase increased (Investigations) | 9 | 1 | 2 | 1
Blood alkaline phosphatase increased (Investigations) | 2 | 0 | 1 | 1
Blood bilirubin increased (Investigations) | 2 | 0 | 1 | 1
Blood cholesterol increased (Investigations) | 3 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 7 | 0 | 1 | 2
Blood lactate dehydrogenase increased (Investigations) | 2 | 0 | 2 | 1
Blood phosphorus decreased (Investigations) | 2 | 0 | 0 | 0
Blood potassium decreased (Investigations) | 2 | 0 | 0 | 0
C-reactive protein increased (Investigations) | 0 | 0 | 0 | 2
Gamma-glutamyltransferase increased (Investigations) | 3 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 1 | 0
Transaminases increased (Investigations) | 0 | 0 | 1 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 3
Decreased appetite (Metabolism and nutrition disorders) | 12 | 0 | 3 | 10
Hypercholesterolaemia (Metabolism and nutrition disorders) | 4 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 3 | 0 | 1 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 3 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 3 | 0 | 1 | 3
Hypocalcaemia (Metabolism and nutrition disorders) | 2 | 0 | 1 | 2
Hypochloraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 0 | 2 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 4 | 1 | 4 | 4
Hypophosphataemia (Metabolism and nutrition disorders) | 3 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 | 0 | 2 | 6
Arthritis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 4
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 3
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 1 | 0 | 1
Sacral pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Dysgeusia (Nervous system disorders) | 3 | 0 | 0 | 3
Headache (Nervous system disorders) | 2 | 0 | 2 | 4
Neuropathy peripheral (Nervous system disorders) | 2 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 1 | 0 | 1 | 0
Anxiety disorder (Psychiatric disorders) | 0 | 0 | 1 | 0
Hallucination (Psychiatric disorders) | 0 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 2 | 0 | 0 | 2
Sleep disorder (Psychiatric disorders) | 0 | 0 | 1 | 0
Micturition urgency (Renal and urinary disorders) | 0 | 0 | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 1 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 3 | 9
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 | 0 | 3 | 9
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 3
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 4
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Nasal ulcer (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 0 | 0 | 2
Rash (Skin and subcutaneous tissue disorders) | 5 | 0 | 1 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 1 | 0 | 2 | 1
Hypotension (Vascular disorders) | 1 | 0 | 1 | 3
Superior vena cava syndrome (Vascular disorders) | 1 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-04-30): https://cdn.clinicaltrials.gov/large-docs/63/NCT04350463/Prot_SAP_000.pdf